CLINICAL TRIAL: NCT02358629
Title: A Prospective, Non-randomized Study to Evaluate the Safety and Performance of the NovaCross™ Microcatheter in Femoropopliteal Chronic Total Occlusion (CTO).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitiloop Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-CPEX-01
Record Dates: First submitted 2015-01-30; First posted 2015-02-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Total Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective, non-randomized (Experimental): use the NovaCross™micro-catheter in respect to providing additional guidewire support that is expected to allow easier crossing of femoropopliteal and infra-popliteal Chronic Total Occlusion (CTO) lesion
  Interventions: Device: NovaCross™ microcatheter

INTERVENTIONS:
Device: NovaCross™ microcatheter — successful delivery, crossing, and retrieval of the investigational device as identified by confirmation of guidewire placement in the distal true lumen confirmed by angiography

SUMMARY:
Trial is to evaluate the safety and performance of the NovaCross™micro-catheter in respect to providing additional guidewire support that is expected to allow easier crossing of femoropopliteal and infra-popliteal Chronic Total Occlusion (CTO) lesion. The procedure will be conducted on a patient diagnosed with a CTO in a peripheral vessel that requires revascularization.

DETAILED DESCRIPTION:
This is an open label, single center, prospective, first in man pilot study in which the investigational device, NitiLoop micro-catheter, will be tested in up to 15 patients with symptomatic peripheral arterial occlusive disease scheduled to undergo CTO in an anterograde approach.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 25-80
2. Patient understands and has signed the study informed consent form.
3. Patient has symptomatic peripheral artery disease (PAD) requiring endovascular revascularization of a CTO, evidenced by angiography, computed tomography or magnetic resonance angiography.
4. Patient has an occluded femoropopliteal or infra popliteal artery
5. Target femoropopliteal or infra-popliteal vessel is ≥ 2.5 mm and ≤5 mm in diameter.
6. Patient has Rutherford-Becker Classification of 2-5.

Exclusion Criteria:

1. Patient unable to give informed consent.
2. Current participation in another study with any investigational drug or device.
3. Patient has a known sensitivity or allergy to contrast materials that cannot be adequately pre-treated.
4. Patient has a known sensitivity or allergy to anti-platelet medications.
5. Patient is pregnant or lactating.
6. Patient has a co-existing disease or medical condition contraindicating percutaneous intervention.
7. Target lesion is in a bypass graft.
8. Target lesion is in a stent (i.e., in-stent restenosis).
9. Patient has had a procedure on the target limb within 7 days.
10. Patient had undergone attempted treatment of the CTO within the prior 3 months (to prevent a guidewire from entering dissection planes created by prior recanalization attempts.
11. Vasculitis and Buerger disease (thrombendarteritis obliterans)
12. Evidence of embolism
13. Peripheral vessel aneurysm

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 30 days
  absence of in-hospital or 30-days Major Adverse Events (MAEs)
Device success is defined as successful delivery, crossing, and retrieval of the investigational device as identified by confirmation of guidewire placement in the distal true lumen confirmed by angiography | in procedure
  Successful femoropopliteal/infra popliteal CTO crossing using the NovaCross™ micro-catheter

CONTACTS AND LOCATIONS:
Overall Officials: Chanan Schneider, Study Chair — Nitiloop Ltd.
Locations (1):
- Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow, Poland